CLINICAL TRIAL: NCT03196596
Title: The Value of Patient-specific Computer Simulation in the Planning of TAVI With the Self-expanding Evolut R Valve
Brief Title: Added Value of Patient-specific Computer Simulation in Transcatheter Aortic Valve Implantation (TAVI)
Acronym: TAVIguide
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: Feops (Industry); Cardialysis B.V. (Industry)
Responsible Party: Principal Investigator, P de Jaegere, MD, PhD, Professor, Erasmus Medical Center
Other Study IDs: TAVIguide
Record Dates: First submitted 2017-06-05; First posted 2017-06-23 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Aortic Valve Stenosis
Keywords: TAVI; Computer simulation
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Computer simulation: Patients in whom a computer simulation model will be obtained based on pre procedural CT
  Interventions: Other: Computer simulation
- Prospective compare group: Patients in whom no computer simulation model will be obtained

INTERVENTIONS:
Other: Computer simulation — In these patients, a computer simulation model will be obtained based on pre procedural CT
  Groups: Computer simulation

SUMMARY:
Transcatheter aortic valve implantation is increasingly used to treat patients with severe aortic stenosis who are at increased risk for surgical aortic valve replacement and is projected to be the preferred treatment modality. As patient selection and operator experience have improved, it is hypothesised that device-host interactions will play a more dominant role in outcome. This, in combination with the increasing number of valve types and sizes, confronts the physician with the dilemma to choose the valve that best fits the individual patient. This necessitates the availability of pre-procedural computer simulation that is based upon the integration of the patient-specific anatomy, the physical and (bio)mechanical properties of the valve and recipient anatomy derived from in-vitro experiments. Patient-specific computer simulation may improve outcome of TAVI by proposing the valve size that best fits the individual patient.

The aim of this study is to assess the added value of patient-specific computer simulation in valve size selection.

ELIGIBILITY:
Inclusion Criteria:

* Native severe aortic valve stenosis
* Planned for TAVI with the Evolut R Valve

Exclusion Criteria:

* Bicuspid aortic valve
* Extensive subannular calcifications
* Non-transfemoral access
* Poor CT quality
* Lack of written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with native severe aortic valve stenosis accepted for TAVI with the self-expanding Evolut R Valve by the local heart team
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2019-01-08 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Decision 1- Valve size decision based on pre TAVI MSCT | an average of 2 days before TAVI, before TAVI and computer simulation
  Valve size decision based on pre TAVI Multislice Computed Tomography (MSCT), which is performed in all patients referred for TAVI in accordance to clinical routine, during the heart team meeting
Decision 2- Valve size decision after knowledge of the computer simulation results | an average of 1 day before TAVI, before TAVI but after computer simulation
  Valve size decision after availability of the results of computer simulation

SECONDARY OUTCOMES:
Decision 3- Change of initial valve size decision during TAVI | an average of 5 minutes after TAVI, directly after TAVI
  Change of valve size decision during TAVI due to computer simulation
Decision 3- Change of initial depth of implantation strategy during TAVI | an average of 5 minutes after TAVI, directly after TAVI
  Change of depth of implantation strategy during TAVI due to computer simulation
Depth of implantation target | an average of 2 days before TAVI, before TAVI and computer simulation
  Initial depth of implantation strategy
Depth of implantation target 2 | an average of 1 day before TAVI, before TAVI but after computer simulation
  Depth of implantation strategy after availability of computer simulation
Aortic regurgitation | an average of 4 days after TAVI, at hospital discharge
  To compare the predicted (simulation) and observed degree of aortic regurgitation (echo post TAVI - Valve Academic Research Consortium (VARC-2) criteria for aortic regurgitation)
Correlation between predicted contact pressure and observed new conduction abnormality | an average of 4 days after TAVI, at hospital discharge
  To compare the predicted maximum contact pressure, contact pressure index and conduction abnormalities with the observed occurrence of new conduction abnormalities after TAVI
MACCE | an average of 4 days after TAVI, at hospital discharge
  To assess the incidence of Major Adverse Cardiovascular and Cerebrovascular Event (MACCE)
Incidence of the aforementioned outcome measures in a prospective group in whom no computer simulation will be perfomed | an average of 4 days after TAVI, at hospital discharge
  To compare the clinical based valve size decision and the angiographic and echocardiographic valve performance, depth of implantation, new conduction disorders and MACCE in a prospectively collected group of patients in whom no computer simulation will be performed

CONTACTS AND LOCATIONS:
Overall Officials: Peter PT de Jaegere, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (5):
- Universitair Ziekenhuis Antwerpen, Edegem, Belgium
- Rigshospitalet, Copenhagen, Denmark
- University Hospital Cologne-Heart Center, Cologne, Germany
- Ospedale di San Raffaele, Milan, Italy
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schultz C, Rodriguez-Olivares R, Bosmans J, Lefevre T, De Santis G, Bruining N, Collas V, Dezutter T, Bosmans B, Rahhab Z, El Faquir N, Watanabe Y, Segers P, Verhegghe B, Chevalier B, van Mieghem N, De Beule M, Mortier P, de Jaegere P. Patient-specific image-based computer simulation for theprediction of valve morphology and calcium displacement after TAVI with the Medtronic CoreValve and the Edwards SAPIEN valve. EuroIntervention. 2016 Jan 22;11(9):1044-52. doi: 10.4244/EIJV11I9A212. PMID 26788707
- [Background] de Jaegere P, De Santis G, Rodriguez-Olivares R, Bosmans J, Bruining N, Dezutter T, Rahhab Z, El Faquir N, Collas V, Bosmans B, Verhegghe B, Ren C, Geleinse M, Schultz C, van Mieghem N, De Beule M, Mortier P. Patient-Specific Computer Modeling to Predict Aortic Regurgitation After Transcatheter Aortic Valve Replacement. JACC Cardiovasc Interv. 2016 Mar 14;9(5):508-12. doi: 10.1016/j.jcin.2016.01.003. No abstract available. PMID 26965945
- [Background] El Faquir N, Ren B, Van Mieghem NM, Bosmans J, de Jaegere PP. Patient-specific computer modelling - its role in the planning of transcatheter aortic valve implantation. Neth Heart J. 2017 Feb;25(2):100-105. doi: 10.1007/s12471-016-0923-6. PMID 27888494